CLINICAL TRIAL: NCT02003625
Title: Non-steroidal Anti-inflammatory Drugs (Meloxicam) to Mobilize Hematopoietic Stem Cells: A Phase II Randomized Trial
Brief Title: Meloxicam vs Placebo for Mobilization
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: The Leukemia and Lymphoma Society (Other)
Responsible Party: Principal Investigator, Bimalangshu Dey, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13-195
Record Dates: First submitted 2013-10-10; First posted 2013-12-06 (Estimated); Results first posted 2020-05-18 (Actual); Last update posted 2020-05-18 (Actual); Status verified 2020-05

CONDITIONS: Non-Hodgkin's Lymphoma; Hodgkin's Lymphoma; Multiple Myeloma; Hematopoietic Stem Cells
Keywords: Non-Hodgkin's lymphoma; Hodgkin's lymphoma; Multiple myeloma; Hematopoietic stem cells
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Hodgkin Disease; Multiple Myeloma | interventions — Meloxicam

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A. GCSF + Placebo (Placebo Comparator): GCSF + Placebo Patients in this group will receive GCSF 10 ug/kg s.c. daily, beginning 4 days prior to the 1st apheresis [days -4, -3, -2, -1] and continued on daily GCSF for a total of 4 apheresis or until ≥ 5 x 10^6 CD34+ cells/kg are collected. They will also receive oral placebo for 5 days on days -6 through -2. Patients will undergo apheresis for 300 minutes to achieve approximately 3 to 4 whole blood volumes processed. This is a standard institutional protocol for autologous HSPC collection at the MGH.
  Interventions: Drug: GCSF; Drug: Placebo
- B. GCSF + meloxicam (Experimental): B. GCSF + meloxicam:
  Patients in this group will be treated with meloxicam and GCSF in an approximate two-day staggered dose schedule as described in our preclinical studies. Meloxicam will be given orally at a dose of 15 mg/day for 5 days (days -6 through -2). GCSF at 10 ug/kg/day subcutaneously will be started on day -4 and continued daily for a total of 4 apheresis or until ≥ 5 x 10^6 CD34+ cells/kg are collected.
  Interventions: Drug: GCSF; Drug: meloxicam

INTERVENTIONS:
Drug: GCSF
Drug: meloxicam
  Arms: B. GCSF + meloxicam
Drug: Placebo
  Arms: A. GCSF + Placebo

SUMMARY:
This research study is evaluating a drug called meloxicam to see if it provides a benefit to people receiving Autologous Hematopoietic Stem Cell Transplantation (AHSCT).

The participant is currently scheduled to receive an AHSCT, which is a procedure that removes blood-forming stem cells (cells from which all blood cells develop) from the body. These stem cells are stored and later given back to the participant by a process called apheresis. This is a standard procedure to treat certain blood diseases such as lymphoma and multiple myeloma. However the use of meloxicam with this procedure is considered investigational.

Meloxicam is a non-steroidal anti-inflammatory drug (NSAID) which is given to decrease fever, swelling and pain that may come with inflammation. It has been approved by the FDA for the treatment of arthritis however it has not been approved for use in people receiving AHSCT.

This study will compare the combination of meloxicam with a drug called G-CSF (also called neupogen), to the combination of G-CSF with an agent that has no medicine (placebo). G-CSF is a substance that causes blood stem cells to change or increase in number when given to people undergoing AHSCT. The researchers would like to learn if giving meloxicam in combination with G-CSF to people before they undergo AHSCT will increase the number of stem cells available in the blood to collect and make the collection process easier.

DETAILED DESCRIPTION:
After the screening procedures confirm that the participant is eligible to participate in the research study:

Because no one knows which of the study options is best, the participant will be "randomized" into one of the study groups:

* G-CSF with meloxicam
* G-CSF with placebo (pills with no medicine)

Randomization means that the participants are put into a group by chance. It is like flipping a coin. Neither the participant nor the research doctor will choose what group the participant will be in. The participant will have an equal chance of being placed in any group.

- Study Drug (meloxicam or placebo): If the participant takes part in this research study, the participant will be given a study drug-dosing diary. The study drug will come as a pill that the participant will take by mouth daily for 5 days, starting 6 days (Day -6) before the participant is scheduled to undergo the first apheresis procedure (Day 0) and continuing until 2 days before apheresis (Day -2). The participant will take meloxicam or placebo for a total of 5 days. The diary will also include special instructions for taking the study drug(s).

-G-CSF: All participants receive G-CSF as an injection under the skin (subcutaneous) in the clinic, daily starting 4 days (Day -4) before the first apheresis procedure (Day 0). The participant will continue to receive G-CSF for 3 days after apheresis.

- Apheresis: The participant may receive up to 4 apheresis procedures, depending on how their body reacts to the stem cell mobilization. The participant will receive either meloxicam or placebo in combination with G-CSF on Days -6 to -2 as described above.

Clinical Exams: While the participant is receiving this procedure, the participant will have regular physical exams and they will be asked specific questions about any problems that they might be having. The participant will also have blood tests every day to look at how their bone marrow is recovering, to give possible transfusional support, and how to see how their liver and kidneys are functioning.

Planned Follow-up: The investigators would like to keep track of the participant's medical condition for the rest of their life. The investigators would like keep track of the participant's medical condition for 6 months after the study to see how they are doing.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet the following criteria on screening examination to be eligible to participate in the study:
* Patients with hematologic malignancies for whom autologous stem cell transplantation is deemed clinically appropriate. Patients participating in this study are patients who are going for their first attempt at stem cell mobilization.
* Non-Hodgkin's lymphoma, or Hodgkin's lymphoma: refractory/relapsed but chemosensitive disease. Patients with CR or PR will be eligible for this protocol.

The designation of PR requires all of the following:

* At least a 50% decrease in sum of the product of the diameters (SPD) of up to six of the largest dominant nodes or nodal masses. These nodes or masses should be selected according to all of the following: they should be clearly measurable in at least 2 perpendicular dimensions; if possible they should be from disparate regions of the body; and they should include mediastinal and retroperitoneal areas of disease whenever these sites are involved.
* No increase should be observed in the size of other nodes, liver, or spleen.
* Splenic and hepatic nodules must regress by ≥ 50% in their SPD or, for single nodules, in the greatest transverse diameter.
* With the exception of splenic and hepatic nodules, involvement of other organs is usually assessable and no measurable disease should be present.
* Bone marrow assessment is irrelevant for determination of a PR if the sample was positive before treatment. However, if positive, the cell type should be specified (eg, large-cell lymphoma or small neoplastic B cells). Patients who achieve a CR by the above criteria, but who have persistent morphologic bone marrow involvement will be considered partial responders. Multiple myeloma in first or second remission. Patients with CR or VGPR will be eligible for this protocol. [VGPR: Serum and urine M-protein detectable by immunofixation only but not on electrophoresis or 90% or greater reduction in serum M-protein plus urine M-protein level <100mg per 24 h]
* Ages 18-75 years
* ECOG performance status of 0, 1, or 2.
* Ability to understand and the willingness to sign a written informed consent
* Patients on NSAIDs will be eligible only when they are off NSAIDs for a month.

Exclusion Criteria:

* Participants who exhibit any of the following conditions at screening will not be eligible for admission into the study.
* Cardiac disease: symptomatic congestive heart failure or RVG or echocardiogram determined left ventricular ejection fraction of < 45%, active angina pectoris, or uncontrolled hypertensionParticipants may not be receiving any other study agents.
* Pulmonary disease: severe chronic obstructive lung disease, or symptomatic restrictive lung disease, or corrected DLCO of < 50% of predicted.
* Renal disease: serum creatinine > 2.0 mg/dl.
* Hepatic disease: SGOT or SGPT > 3 x normal; serum bilirubin >2.0 mg/dl that is not due to Gilbert's syndrome or hemolysis
* Uncontrolled infection.
* Pregnancy or lactation
* Patients with NSAIDs allergies, including patients who have experienced a prior GI bleed due to NSAIDs will be excluded. Patients who have had a recent GI bleed less than 2 weeks ago will be excluded. Patients who are on therapeutic dose anticoagulants will be excluded from this protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-10; Primary Completion 2019-02 (Actual); Study Completion 2019-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bimalangshu Dey, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One patient assigned to the GCSF + placebo arm withdrew consent prior to the start of treatment
Groups:
- A. GCSF + Placebo: GCSF + Placebo Patients in this group will receive GCSF 10 ug/kg s.c. daily, beginning 4 days prior to the 1st apheresis [days -4, -3, -2, -1] and continued on daily GCSF for a total of 4 apheresis or until ≥ 5 x 10^6 CD34+ cells/kg are collected. They will also receive oral placebo for 5 days on days -6 through -2. Patients will undergo apheresis for 300 minutes to achieve approximately 3 to 4 whole blood volumes processed. This is a standard institutional protocol for autologous HSPC collection at the MGH.
  GCSF
  Placebo
- B. GCSF + Meloxicam: B. GCSF + meloxicam:
  Patients in this group will be treated with meloxicam and GCSF in an approximate two-day staggered dose schedule as described in our preclinical studies. Meloxicam will be given orally at a dose of 15 mg/day for 5 days (days -6 through -2). GCSF at 10 ug/kg/day subcutaneously will be started on day -4 and continued daily for a total of 4 apheresis or until ≥ 5 x 10^6 CD34+ cells/kg are collected.
  GCSF
  meloxicam
Period: Overall Study
Arm/Group | A. GCSF + Placebo | B. GCSF + Meloxicam
Started | 15 | 15
Received Transplant | 14 | 12
Completed | 14 | 12
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A. GCSF + Placebo | B. GCSF + Meloxicam | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Median (Full Range); unit: years] | 60 [44 to 74] | 60 [40 to 75] | 60 [40 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 13
  Male | 10 | 7 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 14 | 12 | 26
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 14 | 13 | 27
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Numbers of Circulating CD34+ Cells on the First Day of Apheresis
Description: Numbers of circulating CD34+ cells on the first day of apheresis
Time Frame: 3 days after starting treatment (or 9 days for multiple myeloma patients that received cyclophosphamide)
Measure: Median (Full Range); unit: Cells per microliter
Arm/Group | A. GCSF + Placebo | B. GCSF + Meloxicam
Number analyzed (Participants) | 15 | 15
Cells per microliter | 26 [8.38 to 148.81] | 30.7 [14 to 61.6]

2. Primary Outcome: Number of Apheresis Sessions Required to Collect ≥ 4 x 10^6 CD34+ Cells/kg for Multiple Myeloma Patients and ≥ 2 x 10^6 CD34+ Cells/kg for Lymphoma Patients
Time Frame: Up to 6 days after the start of treatment or up to 12 days for multiple myeloma patients that received cyclophosphamide
Measure: Count of Participants; unit: Participants
Arm/Group | A. GCSF + Placebo | B. GCSF + Meloxicam
Number analyzed (Participants) | 15 | 15
Participants
  1 Session | 4 | 4
  2 Sessions | 6 | 10
  3 Sessions | 4 | 1
  4 Sessions | 1 | 0

3. Primary Outcome: Time to Neutrophil Engraftment After AHSCT
Description: The median to neutrophil engraftment (absolute neutrophil counts above 0.5/mcl for 3 consecutive days) .
Time Frame: Up to 6 months after transplantation ( up to 66-72 days after the start of treatment)
Population: Time to engraftment was only assessed among patients that received transplantation
Measure: Median (Full Range); unit: Days
Arm/Group | A. GCSF + Placebo | B. GCSF + Meloxicam
Number analyzed (Participants) | 14 | 12
Days | 10 [10 to 12] | 10 [9 to 11]

4. Primary Outcome: Time to Platelet Engraftment After AHSCT
Description: The median to platelet engraftment (platelet count above 20,000/mcl for 3 consecutive days)
Time Frame: Up to 6 months after transplantation ( up to 66-72 days after the start of treatment)
Population: Time to engraftment was only assessed among patients that received transplantation
Measure: Median (Full Range); unit: Days
Arm/Group | A. GCSF + Placebo | B. GCSF + Meloxicam
Number analyzed (Participants) | 14 | 12
Days | 18 [11 to 33] | 19 [9 to 23]

5. Secondary Outcome: Number of Patients With Grade 3+ Treatment Related Adverse Events
Description: Adverse events were assessed using Common Terminology Criteria for Adverse Events (CTCAE v4). Related adverse events were defined as adverse events that were deemed to be possibly, probably, or definitely related to study treatment.
Time Frame: Up to 30 days after the last apheresis session (up to 36 days after the start of treatment or 42 days for multiple myeloma patients that received cyclophosphamide)
Measure: Count of Participants; unit: Participants
Arm/Group | A. GCSF + Placebo | B. GCSF + Meloxicam
Number analyzed (Participants) | 15 | 15
Participants | 0 | 0

6. Secondary Outcome: Number of Participants That Received Red Blood Cell and Platelet Transfusions Prior to Engraftment
Time Frame: Up to 6 months after transplantation ( up to 66-72 days after the start of treatment)
Population: Number of transfusions needed were only counted among patients that underwent transplantation
Measure: Count of Participants; unit: Participants
Arm/Group | A. GCSF + Placebo | B. GCSF + Meloxicam
Number analyzed (Participants) | 14 | 12
Participants
  Platelet transfusions | 14 | 9
  Red blood cell transfusions | 6 | 3

7. Secondary Outcome: Number of Patients That Failed to Achieve Stem Cell Mobilization.
Description: The number of patients that did not achieve CD34+ count of ≥ 4 x 10^6 CD34+ cells/kg for multiple myeloma patients or ≥ 2 x 10^6 CD34+ cells/kg for lymphoma patients.
Time Frame: Up to 6 days after the start of treatment or up to 12 days for multiple myeloma patients that received cyclophosphamide
Measure: Count of Participants; unit: Participants
Arm/Group | A. GCSF + Placebo | B. GCSF + Meloxicam
Number analyzed (Participants) | 15 | 15
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 30 days after the last apheresis session (up to 36 days after the start of treatment or 42 days for multiple myeloma patients that received cyclophosphamide)
Description: Only grade 3+ toxicities were recorded for the study
Arm/Group | A. GCSF + Placebo | B. GCSF + Meloxicam
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-28): https://cdn.clinicaltrials.gov/large-docs/25/NCT02003625/Prot_SAP_000.pdf